CLINICAL TRIAL: NCT04931992
Title: Outcome of Patients With CBF and/or NPM1-mutated AML in First Molecular Relapse.
Acronym: MOLAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202100042
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Molecular relapse: Confirmed molecular relapse, without overt cytological relapse
  Interventions: Other: No intervention
- Cytological relapse: Overt cytological relapse, without prior molecular relapse
  Interventions: Other: No intervention
- Persistent responders: No molecular or cytological relapse during follow-up
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Retrospective analysis

SUMMARY:
Despite good initial response, some patients with core binding factor and/or NPM1-mutated AML eventually relapse. Some of these patients can be identified earlier on, before overt cytological relapse, when followed for minimal residual disease. The outcome of patients treated when molecular relapse is confirmed, before overt cytological relapse, is not well known. This multi-center retrospective will therefore study the outcome of these patients and try to specify the role of allogeneic stem cell transplantation in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 61 years
* Diagnosis between 2010 and 2019
* Core binding factor and/or NPM1 acute myeloid leukemia
* First complete remission after induction therapy
* Measurable residual disease measurement after end of consolidation therapy

Exclusion Criteria:

* Acute promyelocytic leukemia
* Allogeneic stem cell transplantation in CR1

Ages: 18 Years to 61 Years | Sex: All
Age Groups: Adult
Study Population: Adult patients < 61 years with CBF and/or NPM1-mutated AML in CR1 after induction therapy who did not receive allogeneic stem transplantation and who were followed for measurable residual disease after completion of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | Up to 5 years

SECONDARY OUTCOMES:
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided